CLINICAL TRIAL: NCT00051467
Title: A Randomized, Phase II/III, Study of TNFerade™ Biologic With 5-FU and Radiation Therapy for First-line Treatment of Unresectable Locally Advanced Pancreatic Cancer
Brief Title: A Study of TNFerade™ Biologic With 5-FU and Radiation Therapy for First-Line Treatment of Unresectable Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GenVec (Industry)
Responsible Party: Paul Fischer, PhD, GenVec
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: GV-001.004; NCT00049647 (obsolete NCT alias)
Record Dates: First submitted 2003-01-10; First posted 2003-01-13 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2011-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

INTERVENTIONS:
Genetic: TNFerade

SUMMARY:
The primary purpose of this study is to assess the safety and effectiveness of TNFerade™ Biologic when administered concurrently with 5-FU and radiation therapy as first-line treatment of unresectable locally advanced pancreatic cancer.

TNFerade™ is a replication deficient adenovirus vector containing the gene for TNF-alpha controlled by a chemoradiation inducible promoter. This allows the expression of TNF-alpha to be greatest in the area receiving radiation. TNF-alpha is a cytokine that has been shown to have potent anti-cancer activities but, due to systemic toxicity, could not be delivered at effective doses. TNFerade™ Biologic is a novel way of selective delivery of TNF-alpha to tumor cells.

TNFerade™ Biologic will be injected during five weekly injection sessions, concomitant with radiation and 5-FU. TNFerade™ Biologic will be administered by direct intratumoral injection using a percutaneous approach (PTA) or endoscopic ultrasound (EUS).

ELIGIBILITY:
Inclusion Criteria

* Age ≥18 years old
* Patients with unresectable, locally advanced adenocarcinoma of the pancreas proven by biopsy or cytology (defined as direct extension to the SMA and/or celiac axis with absence of a fat plane between the low-density tumor and these arterial structures, or loss of patent superior mesenteric-portal vein confluence), who have not received previous treatment for pancreatic cancer. Patients who have been surgically explored and deemed unresectable on that basis are eligible, provided other entry criteria are met
* Informed consent
* Karnofsky performance status = or >70%
* Life expectancy greater than 3 months
* Measurable disease

Exclusion Criteria

* Metastatic (stage IV) disease (including involvement of the colon, adrenals, or kidney, or radiographic evidence of peritoneal seeding)
* Patients with ascites detected by CT, US or MRI
* Patients with bulky celiac adenopathy (i.e., > 2.5 cm)
* Diagnosis of islet cell tumor of the pancreas, lymphoma of the pancreas
* History of other malignancy in the past 2 years except carcinoma in situ of the cervix or bladder, non-melanomatous skin cancer or localized early stage prostate cancer
* Previous chemotherapy or radiation for pancreatic cancer or previous radiation to the target field
* Liver enzymes >3 x ULN (ALT, AST, total bilirubin, alkaline phosphatase)
* Coagulopathy (INR >1.5, PTT ratio >1.5)
* Renal insufficiency (serum creatinine >2.0 mg/dL)
* Significant anemia (e.g. hematocrit <28% or hemoglobin <9 g/dL) (may have RBC transfusion), or thrombocytopenia (platelet count <100,000/µL); or neutropenia (ANC <1500/µL)
* Patients with clinically significant pancreatitis within 12 weeks of treatment
* Pancreatic pseudocyst
* Contraindication to both percutaneous- and endoscopic- guided delivery
* Patients with history of deep venous thrombosis or pulmonary embolus
* Patients with doppler evidence of deep venous thrombosis at screening
* Patients with history of coagulopathy or known thrombophilic disorders
* Patients receiving hormone replacement therapy including oral contraceptives within 2 weeks prior to Day 1.
* Clinical evidence of active infection of any type, including hepatitis B or C virus
* Pregnant or lactating women. It is recommended that both men and women use condoms or another barrier method of birth control for at least 8 weeks following the last administration of TNFerade™ biologic and some form of birth control for at least 1 year
* Experimental medications within the last 4 weeks prior to Day 1
* Surgery within the last 4 weeks prior to Day 1 (if patient was ambulatory within 48 hours of surgery, patient may be considered eligible)
* Chronic systemic corticosteroid use at superphysiologic doses (greater than 10mg prednisone per day or equivalent)
* Significant concurrent medical or psychiatric illness which, in the opinion of the investigator, would interfere with the patient's ability to participate in the trial

Please note that there are additional entry criteria. The study center will determine if you meet all criteria. If you do qualify to participate, study personnel will explain the study and answer any questions you may have. You can decide whether or not you wish to participate but if you do not qualify for this trial, study staff will explain the reasons. Please contact your local center listed below, or call the toll free PACT study line for assistance at 1-888-344-6096

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - UCLA School of Medicine, Division of Hematology-Oncology, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - University of Colorado Health Science Center Facility, Denver, Colorado
  - Georgetown, MedStar Research Institute, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Tampa General Hospital, Tampa, Florida
  - Winship Cancer Center, Emory University, Atlanta, Georgia
  - The Universtiy of Chicago Medical Center, Chicago, Illinois
  - St. James Hospital and Health Centers Comprehensive Cancer Institute, Olympia Fields, Illinois
  - Indiana University Medical Goup, Indianapolis, Indiana
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University, Karmanos Cancer Institute, Detroit, Michigan
  - Research Medical Center, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - Beth Israel Medical Center, BI Cancer Center, New York, New York
  - Leo W. Jenkins Cancer Center, Greenville, North Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Mary Crowley Medical Center, Dallas, Texas
  - Univeristy of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin, Division of Neoplastic Diseases & Related Disorders, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Herman JM, Wild AT, Wang H, Tran PT, Chang KJ, Taylor GE, Donehower RC, Pawlik TM, Ziegler MA, Cai H, Savage DT, Canto MI, Klapman J, Reid T, Shah RJ, Hoffe SE, Rosemurgy A, Wolfgang CL, Laheru DA. Randomized phase III multi-institutional study of TNFerade biologic with fluorouracil and radiotherapy for locally advanced pancreatic cancer: final results. J Clin Oncol. 2013 Mar 1;31(7):886-94. doi: 10.1200/JCO.2012.44.7516. Epub 2013 Jan 22. PMID 23341531